CLINICAL TRIAL: NCT01763346
Title: Beta Cell Restoration Through Fat Mitigation
Acronym: BetaFat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas Buchanan, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BETAFAT; U01DK094430 (NIH); IIT - 000395 (Other Grant/Funding Number: Allergan Corporation)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Prediabetes; Type 2 Diabetes; Obesity
Keywords: type 2 diabetes; prediabetes; obesity; gastric banding; metformin
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Active Comparator): subjects receiving metformin
  Interventions: Drug: Metformin
- gastric banding (Experimental): subjects receiving LAP-BAND
  Interventions: Device: gastric banding

INTERVENTIONS:
Drug: Metformin — metformin 1000 mg bid
  Arms: metformin
Device: gastric banding — LAP-BAND
  Arms: gastric banding

SUMMARY:
Weight loss achieved through gastric banding will be superior to treatment with metformin in preserving or restoring pancreatic beta cell function in people with prediabetes or mild type 2 diabetes.

DETAILED DESCRIPTION:
BetaFat is a 2-arm, unblinded study to compare gastric banding to treatment with metformin over a 24-month period in moderately obese adults with pre- or mild type 2 diabetes. The primary outcome will be change in β-cell compensation for insulin resistance, which the investigators will compare between groups. Secondary analyses will include other potential markers of β-cell health and potential mediators of treatment-specific effects. The main focus will be on mediators related to obesity. Clinically, the project will serve as a test of concept for use of gastric banding relatively early in the spectrum of obesity and β-cell disease. Biologically, the results will provide crucial information on potential mediators of β-cell failure and its arrest or reversal in the context of obesity. Those mediators will guide the development of more effective treatment and monitoring for the β-cell disease that causes type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Prior completion of at least two months in a diet, exercise and lifestyle intervention program within the past two years
2. Fasting plasma glucose >90 mg/dl plus 2-hour glucose ≥140 mg/dl on 75 gm OGTT plus HbA1C ≤7.0%. There is no lower limit for the A1C and no upper limit for the OGTT 2-hour glucose based on prior studies that allow us to identify people with falling β-cell function
3. Age 22-65 years
4. Body mass index (BMI) 30-40 kg/m2
5. For participants with diabetes, known duration <1 year
6. No history of use of antidiabetic medications except during pregnancy

Exclusion Criteria:

1. Contraindications to LapBand(see Appendix 1)
2. Contraindication to MRI (claustrophobia; permanent metal objects such as pacemakers, prostheses, aneurysm clips)
3. Underlying disease(s) likely to (a) limit life span to less than study duration and/or (b) increase risk of intervention outside of the study and/or (c) limit ability to participate in outcomes assessment and/or (d) limit participation
4. An underlying disease known to have important effects on glucose metabolism
5. Active infections
6. Renal disease (serum creatinine ≥1.4 mg/dl for men; ≥1.3 mg/dl for women) or serum potassium abnormality (<3.4 or >5.5 mmol/l)
7. Anemia (hemoglobin <11g/dl in women, <12 g/dl in men) or known coagulopathy
8. Cardiovascular disease, including uncontrolled hypertension and symptomatic congestive heart failure. Participants must be able to safely tolerate administration of fluid/volume challenges during clamp studies.
9. Serum AST >3 times upper limit of normal in local clinical lab
10. Excessive alcohol intake
11. Suboptimally treated thyroid disease
12. Conditions or behaviors likely to affect the conduct of the study

    1. unable or unwilling to give informed consent
    2. unable to adequately communicate with clinic staff
    3. another household member is a participant or staff member
    4. current or anticipated participation in another intervention research project that would interfere with any of the interventions/outcomes
    5. likely to move away from participating clinic in next 2 years
    6. current (or anticipated) pregnancy and lactation.
    7. major psychiatric disorder that, in the opinion of clinic staff, would impede the conduct of the study
    8. weight loss >5% in past three months for any reason except postpartum weight loss.
13. additional conditions may serve as criteria for exclusion at the discretion of the local site

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Buchanan, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] RISE Consortium. Restoring Insulin Secretion (RISE): design of studies of beta-cell preservation in prediabetes and early type 2 diabetes across the life span. Diabetes Care. 2014;37(3):780-8. doi: 10.2337/dc13-1879. Epub 2013 Nov 5. PMID 24194506
- [Result] Xiang AH, Trigo E, Martinez M, Katkhouda N, Beale E, Wang X, Wu J, Chow T, Montgomery C, Nayak KS, Hendee F, Buchanan TA; RISE Consortium; RISE Collaborators. Impact of Gastric Banding Versus Metformin on beta-Cell Function in Adults With Impaired Glucose Tolerance or Mild Type 2 Diabetes. Diabetes Care. 2018 Dec;41(12):2544-2551. doi: 10.2337/dc18-1662. Epub 2018 Oct 3. PMID 30282699
- [Result] RISE Consortium. Metabolic Contrasts Between Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes: I. Observations Using the Hyperglycemic Clamp. Diabetes Care. 2018 Aug;41(8):1696-1706. doi: 10.2337/dc18-0244. Epub 2018 Jun 25. PMID 29941497
- [Derived] Tjaden AH, Edelstein SL, Arslanian S, Barengolts E, Caprio S, Cree-Green M, Lteif A, Mather KJ, Savoye M, Xiang AH, Kahn SE. Reproducibility of Glycemic Measures Among Dysglycemic Youth and Adults in the RISE Study. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1125-e1133. doi: 10.1210/clinem/dgad135. PMID 36938582
- [Derived] Utzschneider KM, Ehrmann DA, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Edelstein SL, Hannon TS, Kahn SE, Kozedub A, Mather KJ, Nadeau KJ, Sam S, Tripputi M, Xiang AH, El Ghormli L; RISE Consortium. Weight loss and beta-cell responses following gastric banding or pharmacotherapy in adults with impaired glucose tolerance or type 2 diabetes: a randomized trial. Obesity (Silver Spring). 2022 Aug;30(8):1579-1588. doi: 10.1002/oby.23475. PMID 35894078
- [Derived] Kahn SE, Edelstein SL, Arslanian SA, Barengolts E, Caprio S, Ehrmann DA, Hannon TS, Marcovina S, Mather KJ, Nadeau KJ, Utzschneider KM, Xiang AH, Buchanan TA; RISE Consortium; Rise Consortium Investigators:. Effect of Medical and Surgical Interventions on alpha-Cell Function in Dysglycemic Youth and Adults in the RISE Study. Diabetes Care. 2021 Sep;44(9):1948-1960. doi: 10.2337/dc21-0461. Epub 2021 Jun 16. PMID 34135015
- [Derived] Kahn SE, Mather KJ, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Ehrmann DA, Hannon TS, Marcovina S, Nadeau KJ, Utzschneider KM, Xiang AH, Edelstein SL; RISE Consortium; Rise Consortium Investigators:. Hyperglucagonemia Does Not Explain the beta-Cell Hyperresponsiveness and Insulin Resistance in Dysglycemic Youth Compared With Adults: Lessons From the RISE Study. Diabetes Care. 2021 Sep;44(9):1961-1969. doi: 10.2337/dc21-0460. Epub 2021 Jun 15. PMID 34131047
- [Derived] Arslanian SA, El Ghormli L, Kim JY, Tjaden AH, Barengolts E, Caprio S, Hannon TS, Mather KJ, Nadeau KJ, Utzschneider KM, Kahn SE; RISE Consortium. OGTT Glucose Response Curves, Insulin Sensitivity, and beta-Cell Function in RISE: Comparison Between Youth and Adults at Randomization and in Response to Interventions to Preserve beta-Cell Function. Diabetes Care. 2021 Mar;44(3):817-825. doi: 10.2337/dc20-2134. Epub 2021 Jan 12. PMID 33436401
- [Derived] RISE Consortium. Obesity and insulin sensitivity effects on cardiovascular risk factors: Comparisons of obese dysglycemic youth and adults. Pediatr Diabetes. 2019 Nov;20(7):849-860. doi: 10.1111/pedi.12883. Epub 2019 Jul 29. PMID 31301210
- [Derived] RISE Consortium. Metabolic Contrasts Between Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes: II. Observations Using the Oral Glucose Tolerance Test. Diabetes Care. 2018 Aug;41(8):1707-1716. doi: 10.2337/dc18-0243. Epub 2018 Jun 25. PMID 29941498
- [Derived] Hannon TS, Kahn SE, Utzschneider KM, Buchanan TA, Nadeau KJ, Zeitler PS, Ehrmann DA, Arslanian SA, Caprio S, Edelstein SL, Savage PJ, Mather KJ; RISE Consortium. Review of methods for measuring beta-cell function: Design considerations from the Restoring Insulin Secretion (RISE) Consortium. Diabetes Obes Metab. 2018 Jan;20(1):14-24. doi: 10.1111/dom.13005. Epub 2017 Jun 22. PMID 28493515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Kaiser Permanente Southern California
Pre-assignment Details: Five participants randomized to metformin and six participants randomized to gastric banding refused to initiate treatment
Period: Overall Study
Arm/Group | Metformin | Gastric Banding
Started | 44 (Five subjects who enrolled in the study refused to initiate metformin therapy, thus did not "start") | 44 (Six subjects randomized to gastric banding refused the banding surgery and, thus, did not "start")
Received Intervention | 39 | 38
Completed | 34 | 36
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Gastric Banding | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 19 | 40
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 31 | 34 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88
Hyperglycemic clamp [Geometric Mean (Inter-Quartile Range); unit: nmol/l adjusted for insulin sensitivity] — data are reported as gemetric mean and 95% confidence interval
  nmol/l adjusted for insulin sensitivity | 3.37 [2.71 to 3.35] | 3.67 [3.28 to 4.1] | 3.52 [2.99 to 3.74]
Oral Glucose Tolerance Test [Mean (Standard Deviation); unit: mmol/l]
  fasting glucose | 6.2 (0.8) | 6.2 (0.7) | 6.2 (0.75)
  2-hour glucose | 10.5 (2.6) | 10.4 (2.7) | 10.45 (2.65)
Body weight [Mean (Standard Deviation); unit: kilograms] | 96.1 (10.9) | 97.5 (12.2) | 96.8 (11.8)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meters squared] | 35.0 (2.9) | 35.7 (2.9) | 35.53 (2.9)
Hemoglobin A1C [Mean (Standard Deviation); unit: percent of hemoglobin] — values are given as standard error and not standard deviation
  percent of hemoglobin | 5.82 (0.06) | 5.92 (0.06) | 5.87 (0.06)

OUTCOME MEASURES:

1. Primary Outcome: Steady State Beta Cell Compensation
Description: mean plasma C-peptide concentration during clamp steady state, adjusted for mean clamp insulin sensitivity
Time Frame: 24 months
Population: Participants completing 24-month hyperglycemic clamp
Measure: Geometric Mean (95% Confidence Interval); unit: (nmol/L) adjusted for M/I
Arm/Group | Metformin | Gastric Banding
Number analyzed (Participants) | 34 | 36
(nmol/L) adjusted for M/I | 3.01 [2.71 to 3.35] | 3.19 [2.88 to 3.53]
Statistical Analysis 1: Comparison: Metformin vs Gastric Banding; We selected a sample size that would allow detection of an effect size of ~0.6 or greater between gastric band and metformin groups for measures of β-cell function after two years, hypothesizing greater function in the gastric band group; Test type: Superiority; p = 0.05, General Linear Models — 35 subjects per group provided 80% power to detect an effect size of 0.59, assuming a 2-sided p=0.05, adjustment for baseline measures using ANCOVA, and correlation of 0.5 between baseline and end-study measures; Differences in primary outcomes between groups at 24-months were compared using general linear models with baseline values included as covariates

2. Other Pre Specified Outcome: Glycemia
Description: fasting and 2-hour OGTT glucose levels
Time Frame: 24 months
Population: participants completing 24 months of interventions
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Metformin | Gastric Banding
Number analyzed (Participants) | 34 | 36
mmol/l
  fasting glucose | 5.95 (0.11) | 5.85 (0.18)
  2-hour glucose | 10.87 (0.57) | 9.92 (0.54)

3. Other Pre Specified Outcome: Glycemia
Description: HbA1C
Time Frame: 24 months
Population: participants completing 24 months of interventions
Measure: Mean (Standard Error); unit: percent of hemoglobin
Arm/Group | Metformin | Gastric Banding
Number analyzed (Participants) | 34 | 36
percent of hemoglobin | 5.84 (0.09) | 5.73 (0.09)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Metformin | Gastric Banding
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/39 | 4/38
Other Adverse Events (participants affected / at risk) | 18/39 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=39) | Gastric Banding (N=38)
gastric band slippage requiring removal (Gastrointestinal disorders) | 0 (0) | 2 (2) — gastric band slippage requireing removal
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
acalcuous cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Requering gall bladder removal
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — requiring fixation, resutling from traffic accident
Gastric sleeve surgery (Gastrointestinal disorders) | 1 (1) | 0 (0) — elective
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=39) | Gastric Banding (N=38)
Port revision (Gastrointestinal disorders) | 0 (0) | 2 (2)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
stomach pain or discomfort (Gastrointestinal disorders) | 11 (11) | 0 (0)
dairrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lack of energy (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT01763346/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT01763346/ICF_001.pdf